CLINICAL TRIAL: NCT02840669
Title: A Study to Characterize the Cardiac Phenotype of Individuals With Friedreich's Ataxia (CARFA Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adverum Biotechnologies, Inc. (Industry)
Collaborators: Adverum Biotechnologies SAS, a wholly owned subsidiary of Adverum Biotechnologies, Inc. (Unknown)
Responsible Party: Sponsor
Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: CM-FA-101
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Friedreich's Ataxia
Keywords: Cardiomyopathy
MeSH Terms: conditions — Friedreich Ataxia; Cardiomyopathies | interventions — Exercise Test

ARMS (2):
- Friedreich's Ataxia (Other)
  Interventions: Procedure: Cardiac magnetic resonance imaging (CMR); Procedure: Exercise-stress test; Procedure: Echocardiography (ECHO); Procedure: Cardiac-related blood studies
- Healthy Volunteers (Controls) (Other)
  Interventions: Procedure: Cardiac magnetic resonance imaging (CMR); Procedure: Exercise-stress test; Procedure: Echocardiography (ECHO); Procedure: Cardiac-related blood studies

INTERVENTIONS:
Procedure: Cardiac magnetic resonance imaging (CMR)
Procedure: Exercise-stress test
Procedure: Echocardiography (ECHO)
Procedure: Cardiac-related blood studies

SUMMARY:
Friedreich's ataxia (FA) is an autosomal recessive disease with an incidence of 1/50,000 in the Caucasian population. The main manifestations of FA are progressive sensory and cerebellar ataxia and cardiomyopathy (CM). It is the most common form of inherited ataxia. A severe CM affects ~60% of FA patients, mostly young adults, and leads to cardiac failure then death. Currently, no therapy can change the course of this severe cardiomyopathy.

This study is designed to characterize the cardiac manifestations of FA using cardiac magnetic resonance (CMR), echocardiography, serum cardiac biomarkers and evaluation of fatigue severity, in the context of the neurological disease.

ELIGIBILITY:
Inclusion Criteria (Friedreich's Ataxia):

* Males and females;
* ≥ 18 years old;
* Willing and able to provide informed consent;
* Definitive diagnosis of FA, based on clinical phenotype and genotype;
* With a hypertrophic cardiomyopathy;
* Ability to complete study assessments.

Exclusion Criteria (Friedreich's Ataxia):

* Symptoms of cardiac failure;
* Moderate to severe atrial or ventricular arrhythmias;
* History of angina pectoris;
* Inability to undergo cardiac MRI;
* Clinical history or evidence of diabetes;
* Abnormal kidney function;
* Females who are pregnant or nursing;
* Receipt of an investigational drug within 30 days or 5 half-lives, or active enrollment in an investigational medication or device study;
* Inability to sit with back support;
* Inability to undergo exercise test;
* Inability to comply with all study requirements;
* Unaffiliated to any French health insurance or equivalent.

Inclusion Criteria (Healthy Volunteers):

* Healthy males and females;
* ≥ 18 years old;
* Willing and able to provide informed consent;
* Age and gender matched to the Friedreich's Ataxia group;
* Ability to complete study assessments.

Exclusion Criteria (Healthy Volunteers):

* Inability to undergo cardiac MRI;
* Clinical history or evidence of diabetes;
* Abnormal kidney function;
* Females who are pregnant or nursing;
* Receipt of an investigational drug within 30 days or 5 half-lives, or active enrollment in an investigational medication or device study;
* Inability to undergo exercise test;
* Inability to comply with all study requirements;
* Unaffiliated to any French health insurance or equivalent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Exercise-stress test | 2 hours
Cardiac magnetic resonance imaging (CMR) | 2 hours
Echocardiogram | 2 hours
Level of cardiac biomarkers in serum | 30 minutes
Fatigue Severity Scale | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Durr, MD, PhD, Principal Investigator — Groupe Hospitalier Pitié-Salpêtrière, APHP
Locations (1):
- Hôpital Pitié-Salpêtrière, AP-HP, Paris, France